CLINICAL TRIAL: NCT01801098
Title: Electrophysiologic HV-interval as a Predicor for Permanent Pacemaker Implantation After Transcatheter Aortic Valve Implantation With a Self-expanding Bioprosthesis
Brief Title: Electrophysiologic HV-interval as a Predicor for Permanent Pacemaker Implantation After TAVI
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Director Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: HV-interval prior TAVI
Record Dates: First submitted 2013-02-06; First posted 2013-02-28 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Symptomatic Aortic Valve Stenosis
Keywords: TAVI; complete AV-block; HV-interval; permanent pacemaker

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The development of a high grade AV-block is a frequent complication associated with transcatheter aortic valve implantation (TAVI). Patients who were suitable for TAVI will be enrolled in this study. The HV-interval will be determined before and immediately after implantation.

The hypothesis is that a prolonged HV-interval is associated with a high rate of complete AV-block following TAVI.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic aortic valve stenosis
* patients screened for TAVI
* written informed consent

Exclusion Criteria:

* unconsciousness, not able to consent
* < 18 years
* permanent pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic aortic valve stenosis screened for TAVI will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Determination of HV interval | Changes in Baseline to 24 hours
  HV-interval will be determined by a 5F quadripolar electrode catheter with a CRD-2 curve configuration. Intracardiac signals will be assessed and determined before and after implantation.

SECONDARY OUTCOMES:
AV-block development after 1 month, 6 months and 12 months | 1 month, 6 months and 12 months

OTHER OUTCOMES:
cardiovascular mortality | 1 month, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Principal Investigator — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Duesseldorf; Marc W. Merx, MD, Principal Investigator — Division of Cardiology, Pulmonary Diseases, Vascular Medicine University Hospital Duesseldorf; Dong-In Shin, MD, Principal Investigator — Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Diseases, Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany